CLINICAL TRIAL: NCT02122185
Title: A Randomized Placebo Controlled Phase II Trial of Metformin in Conjunction With Chemotherapy Followed by Metformin Maintenance Therapy in Advanced Stage Ovarian, Fallopian Tube and Primary Peritoneal Cancer
Brief Title: Metformin and Chemotherapy in Treating Patients With Stage III-IV Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB13-1235; NCI-2014-00860 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB13-1235
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Brenner Tumor; Malignant Ascites; Malignant Pleural Effusion; Ovarian Clear Cell Cystadenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mixed Epithelial Carcinoma; Ovarian Serous Cystadenocarcinoma; Ovarian Undifferentiated Adenocarcinoma; Recurrent Fallopian Tube Cancer; Recurrent Ovarian Epithelial Cancer; Recurrent Ovarian Germ Cell Tumor; Recurrent Primary Peritoneal Cavity Cancer; Stage IIIA Fallopian Tube Cancer; Stage IIIA Ovarian Epithelial Cancer; Stage IIIA Ovarian Germ Cell Tumor; Stage IIIA Primary Peritoneal Cavity Cancer; Stage IIIB Fallopian Tube Cancer; Stage IIIB Ovarian Epithelial Cancer; Stage IIIB Ovarian Germ Cell Tumor; Stage IIIB Primary Peritoneal Cavity Cancer; Stage IIIC Fallopian Tube Cancer; Stage IIIC Ovarian Epithelial Cancer; Stage IIIC Ovarian Germ Cell Tumor; Stage IIIC Primary Peritoneal Cavity Cancer; Stage IV Fallopian Tube Cancer; Stage IV Ovarian Epithelial Cancer; Stage IV Ovarian Germ Cell Tumor; Stage IV Primary Peritoneal Cavity Cancer
MeSH Terms: conditions — Brenner Tumor; Pleural Effusion, Malignant; Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Metformin; Drug Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin plus chemotherapy (Experimental): Patients receive metformin hydrochloride PO BID and standard chemotherapy for 6 -8 cycles. Treatment with metformin hydrochloride continues for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: metformin hydrochloride; Drug: Chemotherapy
- Placebo plus chemotherapy (Placebo Comparator): Patients receive placebo PO BID and standard chemotherapy for 6 -8 cycles. Treatment with placebo continues for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: placebo; Drug: Chemotherapy

INTERVENTIONS:
Drug: metformin hydrochloride — Given PO
  Other Names: Glucophage
  Arms: Metformin plus chemotherapy
Drug: placebo — Given PO
  Other Names: PLCB
  Arms: Placebo plus chemotherapy
Drug: Chemotherapy — Participants will received standard chemotherapy (6-8 cycles). Specific regimen to be given is at the discretion of their treating physician.

SUMMARY:
This randomized phase II trial studies how well metformin hydrochloride and combination chemotherapy works in treating patients with stage III-IV ovarian, fallopian tube, or primary peritoneal cancer. Drugs used in chemotherapy, such as carboplatin, paclitaxel and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Metformin hydrochloride may help carboplatin, paclitaxel and docetaxel work better by making tumor cells more sensitive to the drugs. Studying samples of blood and tissue in the laboratory from patients receiving metformin hydrochloride may help doctors learn more about the effects of metformin hydrochloride on cells. It may also help doctors understand how well patients respond to treatment. Giving metformin hydrochloride together with combination chemotherapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the addition of metformin to standard adjuvant or neoadjuvant chemotherapy plus extended metformin (metformin hydrochloride) beyond standard chemotherapy increases progression free survival when compared to 6 cycles of standard chemotherapy alone in non-diabetic subjects with stage III (with any gross residual disease) or stage IV ovarian, primary peritoneal, or fallopian tube carcinoma.

SECONDARY OBJECTIVES:

I. To determine whether the addition of metformin to standard chemotherapy plus extended metformin beyond standard chemotherapy increases the time to biochemical progression when compared to chemotherapy alone.

II. To compare biochemical (cancer antigen [CA]-125) response rates in the two arms.

III. To describe and compare toxicities in the two arms. IV. To compare overall survival in both arms.

TERTIARY OBJECTIVES:

I. To elucidate metformin's molecular mechanism of action in ovarian, fallopian tube or primary peritoneal cancer by: determining whether metformin's anti-cancer effects are mediated by systemic metabolic changes, a direct effect on tumor cells, or both, and testing the metabolic and proteomic alterations induced in biospecimens from non-diabetic patients prospectively treated with standard chemotherapy in conjunction with metformin compared to placebo.

OUTLINE:

Patients receive a standard chemotherapy regimen at the discretion of the treating physician. Regimens include either paclitaxel intravenously (IV) over 2-3 hours and carboplatin IV over 30-60 minutes on day 1; docetaxel IV over 1 hour on and carboplatin IV over 30-60 minutes on day 1; or paclitaxel IV over 1 hour on days 1, 8, and 15, and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for up to 6 courses. Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive metformin hydrochloride orally (PO) twice daily (BID) and standard chemotherapy regimen as above for 6 courses. Treatment for metformin hydrochloride continues for up to 2 years in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive placebo PO BID and standard chemotherapy regimen as above for 6 courses. Treatment for placebo continues for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

ELIGIBILITY CRITERIA FOR PRE-REGISTRATION

* A reasonable suspicion of ovarian cancer by the treating oncologist is required, evidenced by abdominal carcinomatosis, omental caking, pleural effusions or ascites AND an elevated CA125 > 250 OR CA125:carcinoembryonic antigen (CEA) ratio > 25 OR CA125 =< 250 with no evidence of gastrointestinal (GI) cancer
* Aged 18 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< upper normal institutional limits (except for patients with Gilbert's disease who are eligible despite elevated serum bilirubin level)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.0 × institutional upper limit of normal
* Creatinine =< institutional upper limit of normal (ULN) OR creatinine clearance >= 60 mL/min/1.73 m^2
* Blood glucose =< 126 mg/dL fasting or =< 140 mg/dL nonfasting
* Signed written pre-registration informed consent document

ELIGIBILITY CRITERIA FOR REGISTRATION:

* Histologically confirmed carcinoma consistent with ovarian, fallopian tube, or primary peritoneal carcinoma
* Subjects undergoing primary debulking surgery must have stage III or IV disease and have undergone surgery to include, at a minimum, removal of the uterus, ovaries and fallopian tubes; these patients may be optimally debulked (less than 1 cm residual disease) but must have grossly visible macroscopic residual disease OR be suboptimally debulked
* Subjects for whom neoadjuvant chemotherapy followed by interval cytoreductive surgery is planned must have fine needle aspirate (FNA) or other cytology showing adenocarcinoma OR core biopsies OR surgically directed biopsies showing adenocarcinoma AND CA125 over 250 OR CA125:CEA ratio > 25 OR CA =< 250 with no evidence of GI cancer; they should have presumed stage III or IV disease, generally based on abdominal carcinomatosis, omental caking, pleural effusions or ascites
* Subject and her physician must agree to six cycles or up to 8 cycles of one of the standard of care regimens allowed on this protocol; these regimens (starting dosage) include:

If < 70 years old:

* IV paclitaxel 175 mg/m^2 and carboplatin area under the curve (AUC) 5-6 every 21 days
* IV docetaxel 75 mg/m^2 and carboplatin AUC 5-6 every 21 days
* IV paclitaxel 80 mg/m^2 day 1, 8, and 15 and carboplatin AUC 5-6 day 1 every 21 days

If 70 years or older:

* IV paclitaxel 135 mg/m^2 plus IV carboplatin AUC 5 plus optional G-CSF every 21 days
* IV paclitaxel 60 mg/m^2 day 1, 8, 15 plus IV carboplatin AUC 5 every 21 days (Day 15 paclitaxel optional)
* IV paclitaxel 60 mg/m^2 plus IV carboplatin AUC 2 day 1, 8, and 15 every 21 days

  * ECOG performance status =< 2
  * Leukocytes >= 3,000/mcL
  * absolute neutrophil count >= 1,500/mcL
  * platelets >= 100,000/mcL
  * total bilirubin =< upper normal institutional limits (except for patients with Gilbert's disease who are eligible despite elevated serum bilirubin level)
  * AST(SGOT)/ALT(SGPT) =< 2.0 × institutional upper limit of normal
  * creatinine =< OR institutional ULN OR creatinine clearance >= 60 mL/min/1.73 m^2
  * blood glucose =< 126 mg/dL fasting or =< 140 mg/dL nonfasting
  * women of child-bearing potential must agree to use an effective method of birth control on trial, as the safety of metformin in pregnancy has not been established; an effective method of birth control includes surgical sterilization of woman or her partner, abstinence, or two barrier methods (e.g. condom plus diaphragm); hormonal methods of birth control are not permitted on this study
  * ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

EXCLUSION CRITERIA FOR PRE-REGISTRATION

* Subjects with known diabetes and those taking metformin, sulfonylureas, thiazolidinediones or insulin for any reason
* Patients who are receiving any other investigational agents
* Subjects with comorbidities that would limit their two year survival for reasons other than ovarian cancer
* Concurrent active invasive malignancy or one previously diagnosed with a greater than 30% chance of recurrence in the next two years
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to metformin
* Subjects must not have conditions associated with increased risk of metformin-associated lactic acidosis, including New York Heart Association class III or IV congestive heart failure, history of acidosis of any type, alcoholic liver disease, or habitual intake of 3 or more alcoholic beverages per day
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active major infection, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or nursing women

EXCLUSION CRITERIA FOR REGISTRATION:

* mucinous adenocarcinoma, borderline tumors
* subjects who will undergo intraperitoneal chemotherapy
* subjects receiving neoadjuvant chemotherapy for whom interval debulking surgery (assuming adequate response to therapy) is not planned
* subjects receiving chemotherapy regimens not specified in the inclusion criteria
* subjects should not be participating in other clinical trials of interventions designed to reduce risk of ovarian cancer recurrence or plan to receive off -protocol maintenance therapy (e.g. paclitaxel or bevacizumab)
* subjects with known diabetes, fasting glucose over 126 mg/dL or random glucose over 140 mg/dL and those taking metformin, sulfonylureas, thiazolidenediones or insulin for any reason
* patients who are receiving any other investigational agents
* subjects with comorbidities which would lead to a clinical expectation that they will not survive two years for reasons other than ovarian cancer
* concurrent active invasive malignancy or one previously diagnosed with a greater than 30% chance of recurrence in the next two years
* history of allergic reactions attributed to compounds of similar chemical or biologic composition to metformin
* subjects must not have conditions associated with increased risk of metformin-associated lactic acidosis, including New York Heart Association class III or IV congestive heart failure, history of acidosis of any type, alcoholic liver disease, or habitual intake of 3 or more alcoholic beverages per day
* uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* pregnant or nursing women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-02-25 (Actual); Primary Completion 2027-02-25 (Estimated); Study Completion 2027-02-25 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 and Gynecological Cancer Intergroup (GCIG) criteria | Time from randomization until disease progression or death from any cause, assessed up to 2 years
  Kaplan-Meier curves will be generated and the metformin and placebo groups compared using a logrank test stratified by initial treatment (primary debulking surgery or neoadjuvant therapy). A one-sided alpha level of 0.15 will be used to determine statistical significance. Median PFS and associated 90% confidence interval will be estimated using the method described in Brookmeyer and Crowley. A Cox regression model will also be fit to assess and adjust for the effects of the stratification factor and other baseline covariates (for example, age, ECOG performance status).

SECONDARY OUTCOMES:
Time to biochemical (CA-125) progression using GCIG criteria | Up to 2 years
  Analyzed using Kaplan-Meier curves, stratified logrank test, and Cox regression modeling. CA-125 response rates in the subgroup of patients with elevated CA-125 at entry (i.e., > institutional ULN) will be compared between the two treatment arms using a chi-square test.
Overall survival | Up to 2 years
  Analyzed using Kaplan-Meier curves, stratified logrank test, and Cox regression modeling.
Incidence of adverse events, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 2 years
  Adverse events will be summarized by type, grade, and attribution. Treatment group comparisons will be performed using chi-square or Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Seiko Yamada, Principal Investigator — University of Chicago
Locations (10):
- United States (10):
  - University of Alabama, Birmingham, Alabama
  - Mitchell Cancer Institute - University of South Alabama, Mobile, Alabama
  - City of Hope, Duarte, California
  - NCH Medical Group- Northwest Community Hospital, Arlington Heights, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Mayo Clinic, Rochester, Minnesota